CLINICAL TRIAL: NCT07176884
Title: Non-inferiority of Nurse-performed Versus Interventional Cardiologist-Performed Radial Catheterization in Elective Coronary Angiography: a Single-center, Open-label Randomized Trial.
Acronym: CATHE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal de Compiègne-Noyon (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: CATHE
Record Dates: First submitted 2025-08-28; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Arterial Catheterization; Intensive Care Medicine; Nurse
Keywords: arterial catheterisation by nurse
MeSH Terms: interventions — Nurses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nurse-led intervention (Other): nurse-performed coronary catheterization
  Interventions: Procedure: nurse-performed coronary catheterization
- medical intervention (Other): interventional cardiologist-performed coronary catheterization
  Interventions: Procedure: interventional cardiologist-performed coronary catheterization

INTERVENTIONS:
Procedure: nurse-performed coronary catheterization — nurse-performed coronary catheterization
  Other Names: Nurse
  Arms: nurse-led intervention
Procedure: interventional cardiologist-performed coronary catheterization — interventional cardiologist-performed coronary catheterization.
  Other Names: interventional cardiologist
  Arms: medical intervention

SUMMARY:
Coronary angiography (or coronary arteriography) is a heart examination performed with contrast media to detect and treat coronary stenosis. The procedure involves the insertion of a catheter (a thin flexible tube) into a blood vessel in the groin (femoral) or arm (radial), which is then guided to the heart (cardiac catheterization). In some healthcare institutions, this medical procedure may be performed by a specially trained registered nurse (RN) under the supervision of an interventional cardiologist.

Radial vascular access generally carries a low risk. However, complications such as hematoma, arterial dissection, or secondary occlusion may occur at the puncture site. Fluoroscopy is associated with a certain degree of radiation exposure.

By acquiring skills traditionally within the scope of medical practice, Article 119 of Law No. 2016-41 of January 26, 2016, on the modernization of the healthcare system, created Article L. 4301-1 of the French Public Health Code, introducing the principle of advanced practice for allied health professionals. Since its implementation in July 2018, advanced practice has aimed to achieve two objectives: improving access to care and enhancing patient care pathways, while reducing physicians' workload in targeted conditions.

A local cooperation protocol was submitted to the Regional Health Agency (ARS) on December 14, 2022. Since catheterization is considered a medical act, the submission of such a protocol is mandatory.

This raises the question: Can radial catheterization, as a medical procedure, fall within the scope of advanced nursing practice under the supervision of an interventional cardiologist?

A literature review on nurse-performed cardiac catheterization identified only one publication, in the journal HEART (1997). In this study, nurses from a cardiology department in Oxford, UK, performed the entire coronary angiography procedure. The study demonstrated that a specialized nurse with appropriate baseline experience could be trained to safely perform standard transfemoral cardiac catheterization procedures (including coronary angiography) in low-risk cases. There was no significant difference in performance (complication rates) between the nurse and cardiologists using the same angiographic facility.

The risk of complication in catheterization and angioplasty is estimated at 1 in 1,000 in the literature. The above-mentioned study is the only one addressing our research question and showed no significant difference in complications between nurses and cardiologists. However, the benefit of radial access performed by nursing staff has not been established. Thus, the benefit-risk ratio for participants in our study remains unknown, though the risk is expected to be low, particularly as the procedure performed by the nurse is carried out under medical supervision.

Furthermore, patients will be monitored for at least 8 hours post-procedure, with extended observation depending on clinical evaluation by the treating physician during hospitalization after randomization. Following discharge, patients will be reassessed at 3 months to collect outcome data and follow-up parameters.

Nurses in the cardiology/ICU department are specially trained, with validation of several competencies. Only RNs who have acquired and validated the following eight competencies participate in the CATHE protocol:

Competency 1: Knowledge of cardiology-specific diseases and care.

Competency 2: Management of patients undergoing coronary angiography.

Competency 3: Preparation of the coronary angiography suite.

Competency 4 (part 1/2): Acquisition of knowledge and procedures specific to coronary angiography.

Competency 4 (part 2/2): Acquisition of knowledge and procedures specific to cardiac catheterization activity.

Competency 5: Assistance to the operator during the procedure.

Competency 6: Management of adverse events occurring during the procedure.

Competency 7: Development of professional behavior and skills related to coronary angiography.

Competency 8: Performance of peripheral radial catheter insertion in the coronary angiography suite (within the framework of the local cooperation protocol and the CATHE study).

Each competency is assessed and validated prior to participation.

The primary objective of our study is to demonstrate that in France, an experienced and specially trained registered nurse can safely perform radial catheter insertion under the supervision of an interventional cardiologist. This does not involve femoral catheterization, nor nurse-performed coronary angiography as described in the earlier publication. The study is strictly limited to radial arterial catheterization.

ELIGIBILITY:
Inclusion Criteria:

Male or female

Age ≥ 18 years

Patient has provided written informed consent to participate

Patient scheduled for hospitalization (emergency hospitalizations, e.g., ACS, are excluded) for suspected ischemic heart disease

Radial access

Exclusion Criteria:

Contraindication to coronary angiography: pregnant women (or with laboratory-confirmed pregnancy), parturient, and breastfeeding women will not be included

History of wrist or upper limb arterial surgery

Patient under legal protection, guardianship, or curatorship

Patient not affiliated with a social security system

Access other than the radial artery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1602 (Actual)
Dates: Start 2024-03-14 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2026-03-14 (Estimated)

PRIMARY OUTCOMES:
Success of catheterization on the first attempt | 24 month
  First-attempt catheterization success.
First-attempt catheterization success | 24 month
  First-attempt catheterization success.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Compiègne-Noyon (Unité de Recherche Clinique), Compiègne, France

IPD SHARING:
Plan to Share IPD: Undecided